CLINICAL TRIAL: NCT04389320
Title: Antimalarial and Covid 19 in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Assistant professor, Assiut University
Other Study IDs: covid 19 in RA
Record Dates: First submitted 2020-05-11; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Hydroxychloroquine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid patients receiving hydroxychloroquine: immunoglobulin analyses of covid 19 virus in patients already on hydroxychloroquine and relation to clinical presentation and genetics
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — assess its role in the coarse of covid 19 virus infection

SUMMARY:
The antimalarial agent hydroxychloroquine(HCQ) have been used widely used for the treatment of rheumatoid arthritis and systemic lupus erythematosus. These compounds lead to improvement of clinical and laboratory parameters, but their slow onset of action differ them from glucocorticoids and nonsteroidal antiinflammatory agents.

Among rheumatic diseases, the primary role of HCQ is in the management of articular and skin manifestations of systemic lupus erythematosus (SLE) and the treatment of mild to moderately active rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
The antimalarial agent hydroxychloroquine(HCQ) have been used widely used for the treatment of rheumatoid arthritis and systemic lupus erythematosus.(1) . These compounds lead to improvement of clinical and laboratory parameters, but their slow onset of action differ them from glucocorticoids and nonsteroidal antiinflammatory agents.

Among rheumatic diseases, the primary role of HCQ is in the management of articular and skin manifestations of systemic lupus erythematosus (SLE) and the treatment of mild to moderately active rheumatoid arthritis (RA).

It is difficult to carefully evaluate the onslaught of information that has emerged regarding potential COVID-19 therapies within a few months' time in early 2020. A brief but detailed approach regarding how to evaluate resulting evidence of a study has been presented by F. Perry Wilson, MD, MSCE. By using the example of a case series of patients given hydroxychloroquine plus azithromycin, he provides clinicians with a quick review of critical analyses.

ELIGIBILITY:
Inclusion Criteria:

* rheumatoid arthritis recieving hydroxychloroquine chest infection

Exclusion Criteria:

* patients not used hydroxychloroquine

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: rheumatoid arthritis patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
immunoglobulin mesurement | 1 month
  serum level

CONTACTS AND LOCATIONS:
Locations (1):
- Manal Hassanien, Asyut, Yes, Egypt